CLINICAL TRIAL: NCT02209974
Title: Inhaled Corticosteroids do Not Modify the Systemic Inflammation Induced by Exercise in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Inhaled Corticosteroids in the Systemic Inflammation Induced by Exercise in Patients With COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Son Llatzer (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other); Hospital Son Espases (Other); Spanish Research Center for Respiratory Diseases (Other); Hospital Clinic of Barcelona (Other); Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Principal Investigator, Antonia Fuster, Medicine PhD, Hospital Son Llatzer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC-COPD-2014
Record Dates: First submitted 2014-07-23; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: emphysema; CRP; interleukin-8; dynamic hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Placebo (Placebo Comparator): Inhaled placebo administered to healthy (n=7) and to a half (n=8) of COPD patients
  Interventions: Drug: Inhaled Placebo
- Inhaled corticosteroids (Fluticasone, 0.5 mg) (Experimental): Inhaled corticosteroids administered to the other half (n=8) of COPD patients
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Fluticasone — Administration of inhaled corticosteroids (fluticasone, 0.5 mg) each 12 hours to 8 of the 16 COPD patients versus placebo.
  Other Names: Inhaled Corticosteroids
  Arms: Inhaled corticosteroids (Fluticasone, 0.5 mg)
Drug: Inhaled Placebo
  Arms: Inhaled Placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by pulmonary and systemic inflammation. The effect of inhaled corticosteroids (IC) on inflammation in COPD is controversial.

DETAILED DESCRIPTION:
Physical exercise produces a systemic inflammatory response, both in the healthy individual and in the COPD patient (Rabinovitch et al ERJ 2003; van Helvoort et al Respir Med 2005; Davidson WJ et al. J Appl Physiol). Nevertheless, although it has been described that some of the systemic biomarkers related with COPD (Protein C-Reactive (PCR), interleukin [IL]-8) are associated with a lower tolerance to exercise in COPD patients (García-Río et al. Respir Res 2010), the role of IC on systemic inflammation triggered by exercise in COPD patients remains unknown.

This study explores the hypothesis that the inflammatory response induced by exercise in COPD patients could be with IC treatment.

ELIGIBILITY:
Inclusion Criteria:

* ex-smokers (> 10 packets-year) with moderate-severe COPD patients

Ages: 58 Years to 72 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Differences in response to exercise between healthy and COPD patients | 1 month
  16 COPD patients were compared with 7 healthy, sedentary and nonsmoker controls. All of them carried out an incremental cycle exercise test (ICET) limited by symptoms.
  1 month later, ICET was repeated only by COPD patients.
  Venous blood samples were obtained at rest and during peak exercise.
  Anthropometric, functional and response characteristics to exercise:
  Age, years
  BMI, m2.kg-1
  FEV1/FVC, %
  FEV1, % reference
  Peak charge, watts
  VO2 peak, mL.min-1
  Respiratory quotient
  VE peak, L.min-1
  Fc peak, lpm
  Lactic acid peak, mmol.L-1
  SaO2 basal, %
  SaO2 peak, %

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Fuster, PhD Medicine, Principal Investigator — Hospital Son Llatzer; Jaume Sauleda, PhD Medicine, Study Chair — Hospital Son Espases; Catalina Balaguer, Medicine, Study Chair — Hospital Son Espases; Bernardí Barceló, PhD Medicine, Study Chair — Hospital Son Espases; Angel Rios, Nursing, Study Chair — FISIB Fundació Investigació de les Illes Balears; Amanda Iglesias, Biology, Study Chair — FISIB Fundació Investigació de les Illes Balears; Aina Noguera, Medicine, Study Chair — Hospital Son Espases; Bernat Togores, Medicine, Study Chair — Hospital Son Espases; Alvar Agustí, PhD Medicine, Study Chair — IDIBAPS Hospital Clínic; Ernest Sala-Llinàs, PhD Medicine, Study Chair — Hospital Son Espases
Locations (1):
- Hospital Son Llatzer, Palma de Mallorca, Balearic Islands, Spain